CLINICAL TRIAL: NCT01931345
Title: The SPOT Project: Effect of Counseling Based on Motivational Interviewing Offered in Conjunction With Rapid HIV Testing on the Occurrence of Unprotected Anal Sex and Its Determinants Among Men Who Have Sex With Men (MSM) in Montreal
Brief Title: The SPOT Project : Motivational Interviewing in Conjunction With Rapid HIV Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec a Montréal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jessica Caruso, Research Agent, Université du Québec a Montréal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPOT
Record Dates: First submitted 2013-08-06; First posted 2013-08-29 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: High-risk Sex
Keywords: Rapid HIV testing; MSM; Motivational Interviewing; HIV prevention; HIV/AIDS; At-risk anal intercourse; Randomized trial
MeSH Terms: conditions — Unsafe Sex; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational Interviewing Counseling (Experimental): Counseling developed by the research team based on a motivational interviewing approach
  Interventions: Behavioral: Motivational Interviewing Counseling
- Standard counseling (Active Comparator): Counseling based on Quebec guidelines for rapid HIV testing
  Interventions: Behavioral: Standard counseling

INTERVENTIONS:
Behavioral: Motivational Interviewing Counseling — Counseling developed by the research team based on a motivational interviewing approach
  Arms: Motivational Interviewing Counseling
Behavioral: Standard counseling — Counseling based on Quebec guidelines for rapid HIV testing
  Arms: Standard counseling

SUMMARY:
In 2009, a team of researchers from Montreal, Canada, implemented SPOT, an intervention aimed at reducing HIV transmission among men who have sex with men by offering rapid HIV testing in a community setting. During the first phase, counseling based on Quebec guidelines for rapid HIV testing was offered (standard counseling - SC) and in the second phase, counseling based on motivational interviewing (MIC) was developed and validated. The current phase of the project aims to strengthen the work undertaken during previous phases. The objective of the study is to assess the short and medium term effect of MIC on the occurrence of at-risk anal intercourse and its cognitive determinants. Participants will be randomly assigned to either SC or MIC, and will respond to a baseline questionnaire documenting their sexual behavior and psychosexual profile prior to the intervention at the start of their initial visit (T0). The effect of counseling will be assessed following the intervention at the end of the initial visit (T1), at 3 months after the initial visit (T2) and at 6 months after the initial visit (T3).

DETAILED DESCRIPTION:
In Canada, the prevalence and incidence of HIV remain high among men who have sex with men (MSM). Moreover, epidemiological data show that a significant proportion of transmission can be attributed people who are unaware of their HIV status. To address these challenges, HIV testing has the potential to be a major prevention strategy. Indeed, the combination of testing and treatment (test & treat) is now seen to be one of the most promising strategies in terms of its potential contribution to the eradication of HIV.

To maximize testing among MSM, it has been recommended that services be diversified by offering HIV testing in close proximity to areas where people most at risk for HIV reside and socialize. Rapid HIV testing can also help reduce barriers in access to testing by reaching those most at risk more effectively in non-traditional venues. In addition, testing offers an excellent opportunity and psycho-affective context within which to provide individualized counseling in order to explore preventive practices and testing routines.

Since July 2009, the SPOT project has combined a number of strategies (testing services in close proximity to a residential area; free, anonymous, and rapid HIV testing; individualized preventive counseling) in an original way at an innovative community site located in the heart of Montreal's Gay Village. In the first phase of the study, standard counseling (SC) based on Quebec guidelines for rapid HIV testing was used. During the second, counseling based on a motivational interviewing approach (MIC) was developed and has been provided to participants since May 2011.

Taking advantage of the existing infrastructure, the objective of the current phase of the study is to assess the short and medium term impact of MIC and its cognitive determinants in comparison to SC. The occurrence of at-risk anal intercourse (unprotected anal sex with an HIV-positive partner or partner of unknown HIV status) will be measured at baseline and followed over six months. Four cognitive determinants of at-risk anal sex will also be measured: the importance that participants accord to taking the necessary steps to protect themselves from HIV, perceived personal efficacy in achieving this, intention to do so, and the extent to which participants have planned to do so.

To achieve this objective, a 24 months randomized trial will be implemented SPOT's community site. Participants who present for HIV testing will be randomized between the two conditions, MIC and SC, alternated at a ratio of 1/1 (experimental condition: MIC offered by a community worker; control condition: SC offered by a nurse). Outcome measures will be collected by means of questionnaires. Four measurement times are planned. A baseline questionnaire will be administered prior to pre-test counseling at the start of the initial visit. Outcome measures will be assessed at baseline (T0), and in follow-up questionnaires administered after post-test counseling at the end of the initial visit (T1), at 3 months after the initial visit (T2) and at 6 months after the initial visit (T3). Target enrolment at T0 is 900, for a final sample of 508 participants at T3, representing 254 participants per group (MIC, SC). Mechanisms will be put in place to ensure the integrity of both MIC and SC interventions as well as to retain participants and involve community members in the research process.

In the wake of the recommendations of the Federal Initiative to Address HIV/AIDS in Canada, this study will provide data on the effectiveness of different forms of preventive counseling tailored for use in conjunction with rapid HIV testing. If MIC proves to be effective, the training and clinical supervision offered to intervention staff as well as the tools and quality control procedures developed during the implementation of this approach to counseling will be made available in other settings where testing is offered. Important lessons may also be learned with regards to the organization of services and the benefits and challenges associated with the implementation of this type of HIV prevention infrastructure. Ultimately, this study will contribute to efforts to more effectively combat the HIV epidemic amongst MSM in Canada and reduce the direct and indirect costs associated with HIV in these communities.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18 years of age or older
* Resident of Quebec
* Able to understand French or English
* Unprotected anal sex with a man on at least one occasion in the last 3 years
* HIV-negative or HIV status unknown

Exclusion Criteria:

* Symptoms of fever (over 38°C), headache, muscular pain, fatigue, and/or swollen lymp
* Previously tested at SPOT
* Enrolled as a participant in the IPERGAY study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2013-07; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline occurrence of at-risk anal intercourse at 6 months | Prior to pre-test counseling at the start of participants' initial visit (baseline, T0), after post-test counseling at the end of the initial visit (T1), at 3 months after the initial visit (T2), and at 6 months after the initial visit (T3)
  Occurrence of at-risk anal intercourse will be assessed prior to pre-test counseling at the start of participants' initial visit (baseline, T0), after post-test counseling at the end of the initial visit (T1), at 3 months after the initial visit (T2), and at 6 months after the initial visit (T3).

SECONDARY OUTCOMES:
Change from baseline importance that participants accord to taking the necessary steps to protect themselves from HIV at 6 months | Prior to pre-test counseling at the start of participants' initial visit (baseline, T0), after post-test counseling at the end of the initial visit (T1), at 3 months after the initial visit (T2), and at 6 months after the initial visit (T3)
  Importance that participants accord to taking the necessary steps to protect themselves from HIV will be assessed prior to pre-test counseling at the start of participants' initial visit (baseline, T0), after post-test counseling at the end of the initial visit (T1), at 3 months after the initial visit (T2), and at 6 months after the initial visit (T3).
Change from baseline perceived personal efficacy in protecting themselves from HIV at 6 months | Prior to pre-test counseling at the start of participants' initial visit (baseline, T0), after post-test counseling at the end of the initial visit (T1), at 3 months after the initial visit (T2), and at 6 months after the initial visit (T3)
  Perceived personal efficacy in protecting themselves from HIV will be assessed prior to pre-test counseling at the start of participants' initial visit (baseline, T0), after post-test counseling at the end of the initial visit (T1), at 3 months after the initial visit (T2), and at 6 months after the initial visit (T3)
Change from baseline intention to protect themselves from HIV at 6 months | Prior to pre-test counseling at the start of participants' initial visit (baseline, T0), after post-test counseling at the end of the initial visit (T1), at 3 months after the initial visit (T2), and at 6 months after the initial visit (T3)
  Intention to protect themselves from HIV will be assessed prior to pre-test counseling at the start of participants' initial visit (baseline, T0), after post-test counseling at the end of the initial visit (T1), at 3 months after the initial visit (T2), and at 6 months after the initial visit (T3)
Change from baseline extent to which participants have planned to protect themselves from HIV at 6 months | Prior to pre-test counseling at the start of participants' initial visit (baseline, T0), after post-test counseling at the end of the initial visit (T1), at 3 months after the initial visit (T2), and at 6 months after the initial visit (T3)
  Extent to which participants have planned to protect themselves from HIV will be assessed prior to pre-test counseling at the start of participants' initial visit (baseline, T0), after post-test counseling at the end of the initial visit (T1), at 3 months after the initial visit (T2), and at 6 months after the initial visit (T3)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Otis, Ph.D., Principal Investigator — Université du Québec a Montréal
Locations (1):
- SPOT, 1223-A rue Amherst, Montreal, Quebec, Canada

REFERENCES:
- See also: Our website — http://www.spottestmontreal.com